CLINICAL TRIAL: NCT02179203
Title: Lung Doppler Signals Changes in Response to Cardiac Resynchronization in Heart Failure Patients
Brief Title: Changes in Doppler Signals From the Lung Due to Cardiac Resynchronization in Heart Failure Patients
Status: Completed | Type: Observational
Sponsor: Echosense Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: DOP021
Record Dates: First submitted 2014-06-27; First posted 2014-07-01 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2014-06

CONDITIONS: Change in LDS Signals Due to Cardiac Synchronization Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

SUMMARY:
Study Purpose and Rationale The purpose of this study is to evaluate the lung Doppler signals changes during cardiac resynchronization procedure. As the LDS represent the various mechanical events of cardiac origin it is assumed that they may reflect the relative timing between contraction of the ventricles and atria and thus serve for effective synchronization of these activities.

Aim of the study:

The aim of the study is to assess whether the changes in Lung Doppler Signal (LDS) waves' characteristics will mimic the changes in echocardiographic parameters designed to assess diastolic inflow and systolic flow in patients undergoing Echo-based CRT optimization.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 years or older, who met the indications for cardiac synchronization therapy (CRT) per the ACCF/AHA guidelines, underwent successful system implant for more than 3 months, and were referred to the CRT non-responder clinic at the Ohio State University for CRT- Echo optimization due to absence of clinical improvement in functional class or ejection fraction after the implant per the judgment of the referring physician.

Exclusion Criteria:

1. Chronic atrial fibrillation or new cardiac arrhythmias detected at the time of the visit that are known to affect the response to CRT (Atrial fibrillation, supraventricular tachycardia, ventricular tachycardia, or frequent premature ventricular contractions).
2. CRT device malfunction
3. Inadequate CRT programming that has contributed to lack of response to CRT
4. Coronary sinus lead anatomical or electrical malfunctions at the time of the visit
5. Acute systemic illness that can explain their lack of functional improvement (i.e., anemia, severe electrolyte imbalance, pneumothorax, pericardial effusion, pneumonia)
6. Inability to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with indication for cardiac snchronization therapy
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in Doppler signals before and after CRT | During procedure

CONTACTS AND LOCATIONS:
Overall Officials: Hyesha Hasan, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University 473 West 12th Ave., Columbus, Ohio, United States